CLINICAL TRIAL: NCT00110487
Title: A Double-Blind, Randomized, Placebo-Controlled, Dose-Ranging Study of the Effect of ERB-041 in the Reduction of Symptoms Associated With Endometriosis in Reproductive-Age Women
Brief Title: Study Evaluating ERB-041 in Endometriosis in Reproductive-Age Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3142A2-200
Record Dates: First submitted 2005-05-09; First posted 2005-05-10 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2007-12

CONDITIONS: Endometriosis
Keywords: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — ERB 041

INTERVENTIONS:
Drug: ERB-041

SUMMARY:
The purpose of this investigational study is to determine if a study medication is safe and effective in reducing the symptoms associated with endometriosis; if the study medication reduces the need for pain medication for endometriosis symptoms; and if the study medication improves a participant's ability to carry out daily activities. Qualified participants will receive no cost treatment, which may include study-related examinations, diagnostic procedures including a Pap smear, laboratory testing, and a mammogram (aged 40-45). Qualified participants will also receive study medication at no cost. As a participant, the study volunteer may also experience the satisfaction of knowing she is helping the advancement of women's health care.

ELIGIBILITY:
Inclusion Criteria:

* Surgical diagnosis of endometriosis within 5 years
* Not pregnant and not lactating
* Willing to use non-hormonal contraception, history of regular menstrual cycles

Exclusion Criteria:

* Hysterectomy, surgical treatment for endometriosis within 3 months
* Certain medications for the treatment of endometriosis
* Previous history of a malignancy
* Abnormalities on physical or gyn exams and abnormal lab tests

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200
Dates: Start 2005-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To assess the effects and to compare the safety profile of an investigational
medication on the relief of endometriosis-related symptoms.

SECONDARY OUTCOMES:
Clinical and subject assessment of symptoms related to endometriosis and the
use of analgesia to relieve symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (44):
- United States (44):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Carmichael, California
  - La Jolla, California
  - Redding, California
  - San Diego, California
  - Lakewood, Colorado
  - Aventura, Florida
  - Boynton Beach, Florida
  - Celebration, Florida
  - Clearwater, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Palm Harbor, Florida
  - Alpharetta, Georgia
  - Atlanta, Georgia
  - Arlington Heights, Illinois
  - Champaign, Illinois
  - Chicago, Illinois
  - Oak Brook, Illinois
  - South Bend, Indiana
  - Shreveport, Louisiana
  - Lanham, Maryland
  - Laurel, Maryland
  - Detroit, Michigan
  - Chaska, Minnesota
  - Chesterfield, Missouri
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Charlotte, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Eugene, Oregon
  - Greenville, South Carolina
  - Greer, South Carolina
  - Dallas, Texas
  - Fort Worth, Texas
  - Webster, Texas
  - Sandy City, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Madison, Wisconsin